CLINICAL TRIAL: NCT07067554
Title: An Investigation of the Relationship Between Mothers' Susceptibility to Breastfeeding Myths and Their Motivation to Breastfeed
Brief Title: Breastfeeding Myths and Mothers' Motivation
Status: Recruiting | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Güzin Ünlü Suvari, Principle Investigator, M.Sc. Lecturer, Acibadem University
Other Study IDs: 2025-07/276
Record Dates: First submitted 2025-06-19; First posted 2025-07-16 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Breastfeeding; Maternal Behavior; Health Knowledge, Attitudes, Practice; Motivation
MeSH Terms: conditions — Breast Feeding; Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Breast milk is a unique and irreplaceable source of nutrition for infants, offering protection against many common childhood diseases due to its natural sterility, accessibility, and immune-boosting antibodies. Exclusive breastfeeding for the first six months of life is critical for healthy growth, development, and immune support. Despite global recommendations by WHO and UNICEF, lack of knowledge and inadequate support continue to hinder optimal breastfeeding practices.

One major barrier is the persistence of cultural myths and misconceptions, such as "colostrum should be discarded," or "infants need water after every feeding." These unfounded beliefs may reduce mothers' confidence and lead to early cessation of breastfeeding or premature introduction of complementary foods.

This study aims to examine the relationship between mothers' belief in breastfeeding myths and their motivation to breastfeed. While prior research has explored each factor individually, no known studies have analyzed their interaction.

ELIGIBILITY:
Inclusion Criteria:

* Having an infant aged 0-6 months
* Having breastfed the baby at least once
* Voluntarily agreeing to participate in the study

Exclusion Criteria:

* Having a physical or psychiatric health condition that prevents breastfeeding
* Having had a multiple (twin or more) pregnancy
* Exclusively formula-feeding the baby

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Mothers aged 18 or older with an infant between 0-6 months, meeting eligibility criteria and providing consent.
Sampling Method: Non-Probability Sample
Enrollment: 191 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Demographic, Birth, and Breastfeeding Characteristics of Participants | At baseline (one-time assessment at enrollment)
  Collected using a 25-question Descriptive Information Form developed by the researchers. Includes maternal demographics, pregnancy and birth history, infant characteristics, breastfeeding status, beliefs, and motivational factors.
Belief in Breastfeeding Myths | At baseline (one-time assessment at enrollment)
  Measured using the Breastfeeding Myths Scale developed by Yılmaz Sezer et al. (2024). The scale consists of 30 items in a single dimension. Total scores range from 30 to 150, with higher scores indicating a stronger belief in breastfeeding myths. A cut-off score of 119.50 is used to distinguish between low and high levels of myth belief.
Breastfeeding Motivation | At baseline (one-time assessment at enrollment)
  Breastfeeding motivation was measured using the Breastfeeding Motivation Scale, originally developed by Kestler-Peleg et al. (2015) and adapted into Turkish by Mızrak Şahin et al. (2019). The scale consists of 24 items and assesses five subdimensions: Integrated Regulation, Intrinsic Motivation and Identified Regulation, Introjected Regulation - Social Approval, Introjected Regulation - Social Pressure, and External Regulation - Additional Benefits. Each subdimension score is calculated separately based on the mean of relevant items. Scores range from 1 to 5, with higher scores indicating higher levels of motivation in the respective subdimension.

CONTACTS AND LOCATIONS:
Locations (1):
- Acıbadem University, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be publicly shared due to privacy concerns and the sensitive nature of maternal and infant health information. However, anonymized data may be made available upon reasonable request to the corresponding author after publication of the study results.

REFERENCES:
- [Background] Bulut, M., & Küçük Alemdar, D. (2021). Breastfeeding motivation in mothers of excessive crying infants: A correlation study. Early Child Development and Care, 191(9), 1417-1426. Cohen, J. (1988). Stati
- [Background] Yilmaz Sezer N, Aker MN, Gonenc IM, Topuz S. Development of the Breastfeeding Myths Scale. Breastfeed Med. 2024 Jan;19(1):40-46. doi: 10.1089/bfm.2023.0200. PMID 38241130
- [Background] Mizrak Sahin B, Ozerdogan N, Ozdamar K, Gursoy E. Factors affecting breastfeeding motivation in primiparious mothers: An application of breastfeeding motivation scale based on self-determination theory. Health Care Women Int. 2019 Jun;40(6):637-652. doi: 10.1080/07399332.2018.1526289. Epub 2019 May 29. PMID 31140955
- [Background] Kestler-Peleg M, Shamir-Dardikman M, Hermoni D, Ginzburg K. Breastfeeding motivation and Self-Determination Theory. Soc Sci Med. 2015 Nov;144:19-27. doi: 10.1016/j.socscimed.2015.09.006. Epub 2015 Sep 8. PMID 26372935
- [Background] Chipojola R, Chiu HY, Huda MH, Lin YM, Kuo SY. Effectiveness of theory-based educational interventions on breastfeeding self-efficacy and exclusive breastfeeding: A systematic review and meta-analysis. Int J Nurs Stud. 2020 Sep;109:103675. doi: 10.1016/j.ijnurstu.2020.103675. Epub 2020 Jun 6. PMID 32585447
- [Background] Eram, U. (2017). A review article: Myths, beliefs and malpractices relating to breastfeeding and complementary feeding practices. International Journal of Pharmaceutical Science Invention, 6(6), 14-16.
- [Background] Yildirim Goksen DF, Ozkan S. The effect of online breastfeeding education on breastfeeding motivation: A randomized controlled study. J Pediatr Nurs. 2024 Mar-Apr;75:e42-e48. doi: 10.1016/j.pedn.2023.12.026. Epub 2024 Jan 5. PMID 38182483
- [Background] Koura, H. (2019). Myths about breastfeeding. Al-Azhar Assiut Medical Journal, 17(2), 109-113. https://doi.org/10.4103/AZMJ.AZMJ_47_19
- [Background] Maleki A, Faghihzadeh E, Youseflu S. The Effect of Educational Intervention on Improvement of Breastfeeding Self-Efficacy: A Systematic Review and Meta-Analysis. Obstet Gynecol Int. 2021 Aug 10;2021:5522229. doi: 10.1155/2021/5522229. eCollection 2021. PMID 34422058
- [Background] Marques ES, Cotta RM, Priore SE. [Myths and beliefs surrounding breastfeeding]. Cien Saude Colet. 2011 May;16(5):2461-8. doi: 10.1590/s1413-81232011000500015. Portuguese. PMID 21655719